CLINICAL TRIAL: NCT02585973
Title: Phase Ib Trial of Dose-escalating AZD1775 in Combination With Concurrent Radiation and Cisplatin for Intermediate and High Risk Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Dose-escalating AZD1775 + Concurrent Radiation + Cisplatin for Intermediate/High Risk HNSCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1430
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: AZD1775; Cisplatin; Head and Neck Squamous Cell Carcinoma; HNSCC; Chemoradiotherapy; Radiotherapy; CRT
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — adavosertib; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open label, single-arm, Phase 1b (Other): AZD1775 when added to standard of care concomitant chemotherapy (cisplatin) and radiation
  Interventions: Drug: AZD1775; Drug: Cisplatin; Radiation: Intensity Modulated Radiotherapy Treatments

INTERVENTIONS:
Drug: AZD1775 — AZD1775 given twice daily (BID) for three consecutive days (M-W) concomitantly with standard of care cisplatin and radiation. AZD1775 doses will be escalated in 50 mg increments up to 200 mg BID (M-W) in subsequent cohorts to determine the MTD.
  Other Names: MK-1775 hemihydrate; L001739996-008U
Drug: Cisplatin — 40 mg/m2 IV infused over 1 hour D1 of each week of radiation
  Other Names: cisplatin injection
Radiation: Intensity Modulated Radiotherapy Treatments — Total dose will be 70 Gy at 2Gy/fx, 35 fractions, M to Fri, for 7 weeks
  Other Names: IMRT

SUMMARY:
This open label, single-arm, Phase 1b study is designed to identify the maximum tolerated dose (MTD) using a traditional 3+3 dose escalation design of the WEE-1 inhibitor AZD1775 when added to standard of care chemotherapy (cisplatin) and radiation for the treatment of locally advanced squamous cell cancer of the head and neck (HNSCC).

DETAILED DESCRIPTION:
This open label, single-arm, Phase 1b study is designed to identify the maximum tolerated dose (MTD) using a traditional 3+3 dose escalation design of the WEE-1 inhibitor AZD1775 when added to standard of care chemotherapy (cisplatin) and radiation for the treatment of locally advanced squamous cell cancer of the head and neck (HNSCC). The first cohort will include a starting dose of 50 mg AZD1775 given twice daily (BID) for three consecutive days (M-W) concomitantly with standard of care cisplatin and radiation. AZD1775 doses will be escalated in 50 mg increments up to 200 mg BID (M-W) in subsequent cohorts to determine the MTD.

Up to 24 patients will be enrolled, depending on the rate of dose limiting toxicity (DLT). The investigators plan to characterize the toxicity (and safety) profile of this regimen. Secondary objectives include determination of the recommended phase 2 dose (RP2D; based on safety and other data considerations), objective response rate (ORR) at 12 weeks and progression free survival (PFS). the investigators will also estimate overall survival (OS) if the effective sample size allows. The investigators hypothesize that the investigators' proposed regimen is safe, and will yield an improved ORR and PFS over historical controls. Correlative studies will be performed on archival tissue, and on optional fresh biopsies performed at baseline and mid-treatment. The investigators will explore associations between p53 mutational status at baseline as well as changes in checkpoint markers, with ORR, PFS and OS. Finally, the investigators plan to describe possible changes in QOL, speech and swallowing.

ELIGIBILITY:
Inclusion Criteria:

4.1.1 Age ≥ 18 years of age 4.1.2 ECOG Performance Status ≤ 1 (see section 12.4, Appendix D) 4.1.3 Biopsy proven HNSCC of the oropharynx, larynx, hypopharynx, or oral cavity Stage III-IVB as defined by American Joint Committee on Cancer (AJCC) T0-T4, N0 - N3, M0 4.1.4 4.1.4 Must be considered Intermediate or High Risk

Oropharynx Intermediate risk patients include those who have all of the following:

* HPV/p16 (+) disease, a significant tobacco smoking history (>10 pack years) and N2b-N3 disease OR
* HPV (-) disease, ≤ 10 years of smoking and large tumors (T2-T3)

Oropharynx High risk patients include those who are either:

* HPV (-) with >10 years of smoking, OR
* HPV (-), ≤ 10 years of smoking and T4 disease Oral Cavity, Larynx, Hypopharynx are considered high/intermediate risk (regardless of HPV, p16 or smoking status) 4.1.5 Pre-treatment swallowing evaluation by speech and swallowing therapist, to included a modified barium swallow showing no significant impairment with swallowing oral medications.

4.1.6 Required initial laboratory values:

* HgB ≥ 9.0 g/dL
* ANC≥1500/mm3
* Platelet count ≥ 100,000/mm3
* Serum creatinine ≤1.5 mg/dL and/or calculated creatinine clearance ≥50 mL/min(via Cockroft and Gault, see section 12.2, Appendix B)
* • Bilirubin within normal limits unless patient has Gilbert's disease and then bilirubin ≤ 3 x upper limits of normal (ULN)
* AST and ALT ≤ 3.0 x ULN 4.1.7 No prior definitive surgery for HNSCC 4.1.8 Recommendation to undergo concurrent CRT, as determined by the treating physician, with a curative goal 4.1.9 Women of childbearing potential (WOCBP) should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study. WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year. The two birth control methods can be composed of: two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. Subjects should start using birth control from the screening visit and continue throughout study mandated treatment and for 90 days after the final dose of study drug.

The following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), copper intrauterine device, sponge, or spermicide. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).

4.1.10 Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy and continuing through the last dose of study therapy and for 90 days after the final dose of study drug 4.1.11 Women of childbearing potential (WOCBP) must have negative pregnancy test within 72 hours prior to D1 of treatment 4.1.12 Ability to swallow oral medications 4.1.13 As determined by the enrolling physician or protocol designee, ability of the patient to understand and comply with study procedures for the entire length of the study 4.1.14 Informed consent reviewed and signed

Exclusion Criteria:

4.2.1 Major surgical procedures ≤28 days prior to D1 of AZD1775 or minor surgical procedures ≤7 days; no waiting required following port-a-cath placement 4.2.2 Patients who have received prior radiation therapy for HNSCC 4.2.3 4.2.3 Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 12.3, Appendix C), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.

• ECG ≤450 msec for males and ≤470 msec for females required on screening ECG 4.2.4 AST or ALT ≥3 x ULN (upper limit of normal) and total bilirubin ≥2 x ULN please refer to Appendix 12.5 'Actions required in cases of combined increase of Aminotransferase and Total Bilirubin - Hy's Law', for further instructions 4.2.5 Not deemed a candidate for concurrent CRT for medical reasons, such as uncontrolled infection (including HIV), or uncontrolled diabetes mellitus which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.

4.2.6 Not willing to avoid grapefruit, grapefruit juices, grapefruit hybrids, Seville oranges, pummelos, and exotic citrus fruits from 14 days prior to the dose of study medication, throughout the study, and until 2 weeks after the last dose of AZD1775 due to potential CYP3A4 interaction with the study medication. Orange juice is allowed.

4.2.7 Patient has had prescription or non-prescription drugs or other products (ie, grapefruit juice) known to be moderate to strong inhibitors or inducers of CYP3A4, which cannot be discontinued 14 days before Day 1 of dosing and withheld throughout the study until 14 days after the last dose of AZD1775 (see section 12.5 Appendix E). Co-administration of aprepitant and fosaprepitant during this study is prohibited. Co-treatment with weak inhibitors of CYP3A4 is allowed.

4.2.8 AZD1775 is an inhibitor of breast cancer resistance protein (BCRP). The use of statins including atorvastatin which are substrates for BCRP are therefore prohibited and patients should be moved on to non-BCRP alternatives.

4.2.9 Unable or unwilling to discontinue use of any sensitive CYP3A4 substrates and CYP3A4 substrates with a narrow therapeutic window (see section 12.5, Appendix E) 4.2.10 Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of AZD1775 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection) 4.2.11 Receiving or less than 21 days since receiving any other concurrent cytotoxic, biologic agent(s) or investigational agent 4.2.12 Patients with a "currently active" second malignancy other than non-melanoma skin cancers, non-invasive bladder cancer, "low risk" adenocarcinoma of the prostate and carcinoma in situ of the cervix. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 2 years.

4.2.13 Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 7 weeks
  Estimate maximum tolerated dose of AZD1775 in combination with cisplatin plus radiotherapy

SECONDARY OUTCOMES:
Toxicity profile (Number of patients with adverse events) | 7 weeks
  Number of patients with adverse events
Objective Response Rate | 12 weeks
  Objective Response Rate = partial response (PR) + complete response (CR)

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Sheth, DO, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Lineberger Comprehensive cancer Center website — http://unclineberger.org/
- See also: North Carolina Cancer Hospital website — http://unclineberger.org/about/nccancerhospital
- See also: National Cancer Institute website — http://www.cancer.gov